CLINICAL TRIAL: NCT00199888
Title: Pilot Study of Iodine-124 Labeled Chimeric G250 (124I-cG250) in Presurgical Patients With Renal Masses
Brief Title: Safety Study With the Antibody, cG250, and Isotope, 124-Iodine, to Diagnose Patients With Renal Masses.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LUD2002-003; MSKCC IRB#: 05-004 (Other: MSKCC)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2021-05-14 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Cancer of Kidney; Kidney Cancer; Renal Cancer; Neoplasms, Kidney; Renal Neoplasms; Renal Cell Carcinoma (RCC); Clear Cell Renal Cell Carcinoma
Keywords: Kidney Cancer; Renal Cancer; Neoplasms, Kidney; cG250; antibody; Iodine 124
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 124I-cG250 (Experimental): Patients who were scheduled for surgical resection of renal masses received a single intravenous (IV) dose of 10 mg of 5 milliCurie (mCi) /10 mg 124I-cG250. Patients underwent Positron-Emission Tomography/Computed Tomography (PET/CT) imaging of the whole body on at least 2 occasions: once following injection and once immediately prior to surgical resection. Patients were scheduled for surgical resection of their renal masses on day 8.
  Interventions: Drug: 124-Iodine-cG250 (124I-cG250)

INTERVENTIONS:
Drug: 124-Iodine-cG250 (124I-cG250)

SUMMARY:
The purpose of this study is to see if an antibody (cG250) attached to a radioactive substance (Iodine-124) safely detects clear cell renal cancer in patients with kidney tumors scheduled for surgery.

DETAILED DESCRIPTION:
Antibodies are proteins made by the immune system. They fight things that the body sees as foreign, such as bacteria and viruses. The body can also see cancer cells as foreign. When the body sees a foreign invader, it sends out antibodies that tag the invader. Once this happens, the immune system can work to destroy whatever the antibody has tagged.

Monoclonal antibodies are antibodies that can be made in the lab. They tag a portion of a cancer cell. Early monoclonal antibodies were made from antibodies grown in mice. They caused an antibody response in humans after one dose. Now they are more like human antibodies, and thus, do not produce the same reactions on repeated doses. These are called chimeric antibodies. The antibody we will use in this study is called chimeric G250 (cG250).

Recent research has shown that some antibodies can attach themselves to cancer cells, and that they bind to very few normal cells. This could help cancer treatment in two ways. One is that the body's own immune system might work to destroy tagged cancer cells. The other is that we can attach chemotherapy drugs or radioactive chemicals to the antibodies. These can then deliver treatment when the antibodies attach to the cancer cells.

This study is being done to test the tagging ability of cG250 to cancer cells. After you receive cG250, you will have a scan. The picture the scan produces will show where the antibody has collected inside the body. From this, it is possible to measure how well cG250 can detect kidney cancer. This is NOT a treatment for renal cancer. After your surgery, we will examine the tumor and other tissue to see how much of the antibody has attached to the tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of a renal mass.
2. Scheduled for surgical resection of renal mass.
3. Expected survival of at least 3 months.
4. Karnofsky performance scale ≥70.
5. The following laboratory results should be within the following limits within the last 4 weeks prior to study day 1:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 10E9/L
   * Platelet count ≥ 100 x 10E9/L
   * Serum bilirubin ≤ 2.0 mg/dL
   * Aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal (ULN)
   * Alanine aminotransferase (ALT) ≤ 2.5 x ULN
   * Serum creatinine ≤ 2.0 mg/dL
6. Pregnancy Test to be performed on female patients of childbearing potential within 24-48 hours before administration of radioactive material.
7. Recovered from toxicity of any prior therapy.
8. Able and willing to give valid written informed consent.

Exclusion Criteria:

1. Intercurrent medical condition that may limit the amount of antibody to be administered.
2. Intercurrent medical condition that renders the patient ineligible for surgery.
3. New York Heart Association Class III/IV cardiac disease.
4. History of autoimmune hepatitis.
5. Chemotherapy, radiotherapy, or immunotherapy within 4 weeks prior to the first cG250 dose.
6. Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study.
7. Lack of availability for immunological and clinical follow-up assessments.
8. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to enrollment.
9. Women who are pregnant or breastfeeding.
10. Allergy to iodine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-06 (Actual); Primary Completion 2006-03 (Actual); Study Completion 2009-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chaitanya R Divgi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Pual Russo, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Divgi CR, Pandit-Taskar N, Jungbluth AA, Reuter VE, Gonen M, Ruan S, Pierre C, Nagel A, Pryma DA, Humm J, Larson SM, Old LJ, Russo P. Preoperative characterisation of clear-cell renal carcinoma using iodine-124-labelled antibody chimeric G250 (124I-cG250) and PET in patients with renal masses: a phase I trial. Lancet Oncol. 2007 Apr;8(4):304-10. doi: 10.1016/S1470-2045(07)70044-X. PMID 17395103

RESULTS

PARTICIPANT FLOW:
Groups:
- 124-Iodine-cG250 (124I-cG250): Patients who were scheduled for surgical resection of renal masses received a single intravenous (IV) dose of 10 mg of 5 milliCurie (mCi)/10 mg 124I-cG250. Patients underwent Positron-Emission Tomography/Computed Tomography (PET/CT) imaging of the whole body on at least 2 occasions: once following injection and once prior to surgical resection. Patients were scheduled for surgical resection of their renal masses on day 8.
Period: Overall Study
Arm/Group | 124-Iodine-cG250 (124I-cG250)
Started | 26
Completed | 25
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: All patients who enrolled in the study and received 124-Iodine-cG250 (124I-cG250).
Groups:
- 124-Iodine-cG250 (124I-cG250): Patients who were scheduled for surgical resection of renal masses received a single intravenous (IV) dose of 10 mg of 5 mCi/10 mg 124I-cG250. Patients underwent PET/CT imaging of the whole body on at least 2 occasions: once following injection and once prior to surgical resection. Patients were scheduled for surgical resection of their renal masses on day 8.
Arm/Group | 124-Iodine-cG250 (124I-cG250)
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Positive Predictive Value (PPV) of 124I-cG250 Based on Positron-Emission Tomography/Computed Tomography (PET/CT) Imaging in the Detection of Clear Cell Renal Cell Carcinoma (RCC) Compared to Pathology of Tumor Mass at Surgical Resection.
Description: Patients were listed as PET-positive based on a tumor to nontumor radioactive uptake ratio of > 3 and PET-negative if less than or equal to 3.
  The resected renal mass (tumor) was subjected to pathological evaluation, and a diagnosis of clear cell RCC or non-clear cell RCC was made.
  PPV is the proportion of patients with a positive PET scan who actually have the disease based on pathology. Patients who have a positive PET scan on imaging and clear cell RCC on pathology will be considered true-positives. Patients who have negative PET scans on imaging and non-clear cell RCC on pathology will be considered true-negatives. Patients with positive PET scans on imaging and non-clear cell RCC on pathology will be considered false positives and those with clear cell RCC on pathology but negative PET scans on imaging will be considered false negatives.
Time Frame: 8 days
Population: All patients who enrolled in the study, received 124I-cG250, had evaluable PET scans, had tissue samples analyzed and were PET-positive. One patient was excluded because the immunoreactivity of the 124I-cG250 administered was < 25% and considered immunologically inactive. Fifteen patients were PET-positive.
Measure: Number (95% Confidence Interval); unit: percent of PET-positive patients
Groups:
- 124-Iodine-cG250 (124I-cG250): Patients who were scheduled for surgical resection of renal masses and received a single intravenous (IV) dose of 10 mg of 5 mCi/10 mg 124I-cG250. Patients underwent PET/CT imaging of the whole body on at least 2 occasions: once following injection and once prior to surgical resection on day 8.
Arm/Group | 124-Iodine-cG250 (124I-cG250)
Number analyzed (Participants) | 15
percent of PET-positive patients | 100 [78 to 100]

2. Secondary Outcome: Negative Predictive Value (NPV) of 124I-cG250 Based on Positron-Emission Tomography/Computed Tomography (PET/CT) Imaging in the Detection of Clear Cell Renal Cell Carcinoma (RCC) Compared to Pathology of Tumor Mass at Surgical Resection.
Description: Patients were listed as PET-positive based on a tumor to nontumor radioactive uptake ratio of > 3 and PET-negative if less than or equal to 3.
  The resected renal mass (tumor) was subjected to pathological evaluation, and a diagnosis of clear cell RCC or non-clear cell RCC was made.
  NPV is the ratio of participants who do not have clear cell RCC to all those who had negative PET scans.
  Patients who have a positive PET scan on imaging and clear cell RCC on pathology will be considered true-positives. Patients who have a negative PET scan on imaging and do not have clear cell RCC on pathology will be considered true-negatives. Patients with a positive PET scan on imaging and do not have clear cell RCC on pathology will be considered false positives and those with clear cell RCC on pathology but negative PET scans on imaging will be considered false negatives.
Time Frame: 8 days
Population: All patients who enrolled in the study, received 124-Iodine-cG250 (124I-cG250), had evaluable PET/CT scans, tissue samples taken and were PET-negative. One patient was excluded because the immunoreactivity of the 124I-cG250 administered was < 25% and considered immunologically inactive. Ten patients were PET-negative.
Measure: Number (95% Confidence Interval); unit: percent of PET-negative patients
Arm/Group | 124-Iodine-cG250 (124I-cG250)
Number analyzed (Participants) | 10
percent of PET-negative patients | 90 [55 to 100]

3. Secondary Outcome: Sensitivity of 124I-cG250 Based on Positron-Emission Tomography/Computed Tomography (PET/CT) Imaging in the Detection of Clear Cell Renal Cell Carcinoma (RCC) Compared to Pathology of Tumor Mass at Surgical Resection.
Description: Patients were listed as PET-positive based on a tumor to nontumor radioactive uptake ratio of > 3 and PET-negative if less than or equal to 3.
  The resected renal mass (tumor) was subjected to pathological evaluation, and a diagnosis of clear cell RCC or non-clear cell RCC was made.
  Sensitivity is defined as the ratio of the proportion of the patients who have clear cell RCC based on pathology and whose PET scans are positive over the number of patients with clear cell RCC. Patients who have a positive PET scan on imaging and clear cell RCC on pathology will be considered true-positives. Patients who have a negative PET scan on imaging and do not have clear cell RCC on pathology will be considered true-negatives. Patients with a positive PET scan on imaging and do not have clear cell RCC on pathology will be considered false positives and those with clear cell RCC on pathology but negative PET scans on imaging will be considered false negatives.
Time Frame: 8 days
Population: All patients who enrolled in the study, received 124-Iodine-cG250 (124I-cG250), had evaluable PET/CT scans, tissue samples taken and had a pathological diagnosis of clear cell renal cell carcinoma. One patient was excluded because the immunoreactivity of the 124I-cG250 administered was < 25% and considered immunologically inactive. Sixteen patients had clear cell renal cell carcinoma.
Measure: Number (95% Confidence Interval); unit: percent of clear cell RCC patients
Arm/Group | 124-Iodine-cG250 (124I-cG250)
Number analyzed (Participants) | 16
percent of clear cell RCC patients | 94 [70 to 100]

4. Secondary Outcome: Specificity of 124I-cG250 Based on Positron-Emission Tomography/Computed Tomography (PET/CT) Imaging in the Detection of Clear Cell Renal Cell Carcinoma (RCC) Compared to Pathology of Tumor Mass at Surgical Resection.
Description: Patients were listed as PET-positive based on a tumor to nontumor radioactive uptake ratio of > 3 and PET-negative if less than or equal to 3.
  The resected renal mass (tumor) was subjected to pathological evaluation, and a diagnosis of clear cell RCC or non-clear cell RCC was made.
  Specificity is defined as the number of patients with non-clear cell RCC correctly classified divided by all non-clear cell RCC patients.
  Patients who have a positive PET scan on imaging and clear cell RCC on pathology will be considered a true-positive. Patients who have a negative PET scan on imaging and do not have clear cell RCC on pathology will be considered true negatives. Patients with a positive PET scan on imaging and do not have clear cell RCC on pathology will be considered false positives and those with clear cell RCC on pathology but negative PET scans on imaging will be considered false negatives.
Time Frame: 8 days
Population: All patients who enrolled in the study, received 124-Iodine-cG250 (124I-cG250), had evaluable PET/CT scans, tissue samples taken and did not have clear cell renal cell carcinoma. One patient was excluded because the immunoreactivity of the 124I-cG250 administered was < 25% and considered immunologically inactive. Nine patients did not have clear cell RCC.
Measure: Number (95% Confidence Interval); unit: percent of non clear cell RCC patients
Arm/Group | 124-Iodine-cG250 (124I-cG250)
Number analyzed (Participants) | 9
percent of non clear cell RCC patients | 100 [66 to 100]

ADVERSE EVENTS:
Time Frame: 35 days
Description: Patients were monitored for adverse events following administration of 124I-cG250. Toxicity was evaluated according to the National Cancer Institute Common Toxicity Criteria (CTC) Scale Version 3.0.
Groups:
- 124-Iodine-cG250 (124I-cG250): Patients who were scheduled for surgical resection of renal masses received a single intravenous (IV) dose of 10 mg of 5 mCi/10 mg 124I-cG250. Patients underwent PET/CT imaging of the whole body on at least 2 occasions: once following injection and once prior to surgical resection. Patients were scheduled for surgical resection of their renal masses 8 days after infusion.
Arm/Group | 124-Iodine-cG250 (124I-cG250)
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 1/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 124-Iodine-cG250 (124I-cG250) (N=26)
Abdominal pain (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 124-Iodine-cG250 (124I-cG250) (N=26)
Lymphopenia (Blood and lymphatic system disorders) | 6
Hyperbilirubinemia (Hepatobiliary disorders) | 9
Haemoglobin decreased (Investigations) | 26
Aspartate aminotransferase increased (Investigations) | 15
Blood creatinine increased (Investigations) | 14
Alanine aminotransferase increased (Investigations) | 11
Platelet count decreased (Investigations) | 9
International normalised ratio increased (Investigations) | 5
Activated partial thromboplastin time prolonged (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Blood bicarbonate decreased (Investigations) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 25
Hyperglycaemia (Metabolism and nutrition disorders) | 24
Hypokalaemia (Metabolism and nutrition disorders) | 5
Hyponatraemia (Metabolism and nutrition disorders) | 5
Hypernatraemia (Metabolism and nutrition disorders) | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No